CLINICAL TRIAL: NCT07242443
Title: A Randomized Controlled Trial Comparing Tegoprazan 50 mg BID Combined With Amoxicillin 1 g TID Versus Tegoprazan 50 mg BID Combined With Amoxicillin 1.5 g BID for the Eradication of Helicobacter Pylori
Brief Title: Tegoprazan Plus Amoxicillin BID vs TID Regimens for H. Pylori Eradication（Frequency Adjusted Same-dose Therapy for H. Pylori）
Acronym: FAST-HP
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: First People's Hospital of Hangzhou (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HP-TGZ-AMO-3g-FrequencyStudy; BCF-LX-XH-20221014-26 (Other Grant/Funding Number: Bethune Charitable Foundation)
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: HELICOBACTER PYLORI INFECTIONS
Keywords: Helicobacter pylori; H. pylori; Amoxicillin; Tegoprazan; Dual Therapy; BID Dosing; TID Dosing; Fixed-Dose Regimen; P-CAB; Frequency Comparison; Antibiotic Regimen Optimization
MeSH Terms: interventions — tegoprazan; Amoxicillin; BID protein, human

STUDY DESIGN:
Intervention Model Description: This is a randomized, two-arm, parallel-group study in which participants are allocated in a 1:1 ratio to receive tegoprazan plus amoxicillin 1 g TID or tegoprazan plus amoxicillin 1.5 g BID for 14 days.
Masking Description: This is an open-label trial. Masking is not feasible because the two study arms use different dosing frequencies (BID vs TID), which cannot be blinded to participants or study personnel.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tegoprazan 50 mg BID + Amoxicillin 1 g TID (Active Comparator): Participants in this arm will receive tegoprazan 50 mg orally twice daily (BID) in combination with amoxicillin 1 gram orally three times daily (TID) for 14 days. This regimen represents the standard dual therapy dosing schedule for Helicobacter pylori eradication.
  Interventions: Drug: Tegoprazan 50 mg; Drug: Amoxicillin 1 g TID
- Tegoprazan 50 mg BID + Amoxicillin 1.5 g BID (Experimental): Participants in this arm will receive tegoprazan 50 mg orally twice daily (BID) in combination with amoxicillin 1.5 grams orally twice daily (BID) for 14 days. This regimen delivers the same total daily dose of amoxicillin (3 grams) as the standard therapy but uses a reduced dosing frequency to evaluate whether a BID schedule can improve convenience, adherence, and eradication outcomes.
  Interventions: Drug: Tegoprazan 50 mg; Drug: Amoxicillin 1.5 g BID

INTERVENTIONS:
Drug: Tegoprazan 50 mg — Tegoprazan 50 mg administered orally twice daily (BID) for 14 days.
Drug: Amoxicillin 1 g TID — Amoxicillin 1 gram administered orally three times daily (TID) for 14 days.
  Arms: Tegoprazan 50 mg BID + Amoxicillin 1 g TID
Drug: Amoxicillin 1.5 g BID — Amoxicillin 1.5 grams administered orally twice daily (BID) for 14 days.
  Arms: Tegoprazan 50 mg BID + Amoxicillin 1.5 g BID

SUMMARY:
This study is designed to evaluate two different tegoprazan-based dual therapy regimens for the treatment of Helicobacter pylori (H. pylori) infection. All participants will receive tegoprazan 50 mg twice daily for 14 days, combined with one of two amoxicillin dosing schedules that contain the same total daily dose of 3 grams of amoxicillin.

One group will receive amoxicillin 1 gram three times daily (TID), which is the standard regimen. The other group will receive amoxicillin 1.5 grams twice daily (BID), an alternative schedule that may improve convenience and treatment adherence while maintaining the same total daily antibiotic amount.

A total of 240 adults with confirmed H. pylori infection will be randomly assigned to one of the two treatment groups. The main goal of the study is to compare the H. pylori eradication rates between the two regimens. Eradication will be assessed 4 to 8 weeks after completing therapy using a ¹³C-urea breath test. Safety, tolerability, and medication adherence will also be monitored.

DETAILED DESCRIPTION:
Helicobacter pylori (H. pylori) infection is a common and clinically important condition associated with peptic ulcer disease, gastric mucosa-associated lymphoid tissue lymphoma, and gastric cancer. Effective eradication remains essential for reducing long-term complications. Traditional proton pump inhibitor (PPI)-based regimens have faced challenges due to rising antibiotic resistance and suboptimal acid suppression.

Tegoprazan is a potassium-competitive acid blocker (P-CAB) that provides rapid, potent, and sustained gastric acid inhibition, which may enhance the effectiveness of amoxicillin-based dual therapy. Amoxicillin resistance remains low in many regions, and its efficacy is closely related to maintaining intragastric pH levels that support bacterial replication.

The standard tegoprazan dual therapy uses amoxicillin 1 gram three times daily (TID). However, TID dosing may affect patient adherence, which can influence eradication outcomes. This study explores an alternative regimen: amoxicillin 1.5 grams twice daily (BID). The two regimens deliver the same total daily dose of 3 grams of amoxicillin, but the BID schedule may improve convenience and medication compliance while maintaining appropriate pharmacodynamic exposure.

This randomized, controlled clinical trial is designed to compare the eradication efficacy, safety, and tolerability of these two dosing strategies in adults with confirmed H. pylori infection. By evaluating whether a simplified BID regimen can achieve non-inferior or superior eradication rates compared with the standard TID regimen, the study aims to provide evidence that may support more convenient dual therapy options for H. pylori management.

ELIGIBILITY:
Inclusion Criteria:

- 1.Adults aged 18 to 70 years. 2.Confirmed Helicobacter pylori infection by ¹³C-urea breath test, stool antigen test, or gastric biopsy.

3.Able to provide written informed consent. 4.Willing and able to comply with all study procedures, including follow-up testing 4-8 weeks after treatment.

Exclusion Criteria:

* 1.Known allergy or hypersensitivity to tegoprazan, amoxicillin, or any β-lactam antibiotics.

  2.Use of antibiotics, proton pump inhibitors (PPIs), bismuth-containing agents, or potassium-competitive acid blockers within 4 weeks before screening.

  3.Severe hepatic impairment (ALT or AST > 3 × upper limit of normal). 4.Severe renal impairment (estimated glomerular filtration rate < 30 mL/min/1.73 m²).

  5.Pregnant or breastfeeding women. 6.History of gastric surgery or conditions that may affect gastrointestinal absorption.

  7.Participation in another clinical trial within the past 30 days. 8.Any condition that, in the investigator's judgment, would make the participant unsuitable for the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-11-20 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
H. pylori Eradication Rate | 4 to 8 weeks after completion of therapy
  Eradication of Helicobacter pylori infection confirmed by a negative ¹³C-urea breath test performed 4 to 8 weeks after the end of the 14-day treatment regimen.

SECONDARY OUTCOMES:
Incidence of Adverse Events | From Day 1 to Day 14 (treatment period)
  The number and proportion of participants reporting any adverse events during the 14-day treatment period, assessed by patient report, clinical evaluation, and laboratory findings.
Incidence of Serious Adverse Events (SAEs) | From Day 1 to study completion (approximately 8-10 weeks)
  Serious adverse events, defined according to standard regulatory criteria (life-threatening events, hospitalization, significant disability, or other medically significant events).
Medication Adherence Rate | Day 1 to Day 14
  Adherence assessed by pill count and participant self-report. Adherence will be expressed as the percentage of prescribed doses actually taken during the 14-day treatment period.
Change in Gastrointestinal Symptom Scores | Baseline to Day 14
  Improvement in gastrointestinal symptoms (such as epigastric discomfort, bloating, nausea), assessed using a standardized symptom questionnaire. Higher scores indicate more severe symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Hangzhou First People's Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided
The plan for sharing individual participant data (IPD) has not yet been determined. A decision regarding IPD sharing will be made after the completion of the study and review of institutional policies and publication requirements.